CLINICAL TRIAL: NCT04366596
Title: Comparison of Drug-eluting Balloon and Plain Balloon for Treatment of Non-atherosclerotic Renal Artery Stenosis: a Randomized Controlled Study
Brief Title: Drug-eluting Balloon for Treatment of Non-atherosclerotic Renal Artery Stenosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-2133
Record Dates: First submitted 2020-03-03; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2019-09

CONDITIONS: Hypertension, Renovascular
Keywords: Renal Artery Obstruction; Takayasu Arteritis; Fibromuscular Dysplasia
MeSH Terms: conditions — Hypertension, Renovascular; Renal Artery Obstruction; Takayasu Arteritis; Fibromuscular Dysplasia | interventions — Angioplasty

STUDY DESIGN:
Intervention Model Description: intervention group: treated with drug eluting balloon control group :treated with plain old balloon
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients are randomly allocated into intervention and control group. The investigator and outcomes assessor only kwow the random number. The participants will not be told the exact group that they were allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEB group (Experimental): angioplasty with paclitaxel eluting balloon
  Interventions: Device: Angioplasty with paclitaxel eluting balloon
- POB group (Placebo Comparator): Angioplasty with plain old balloon
  Interventions: Device: Angioplasty with plain old balloon

INTERVENTIONS:
Device: Angioplasty with paclitaxel eluting balloon — The patients will be treated with renal artery angioplasty using paclitaxel eluting balloon
  Arms: DEB group
Device: Angioplasty with plain old balloon — Angioplasty with plain old balloon
  Arms: POB group

SUMMARY:
Efficacy of drug eluting balloon(DEB) for non-atherosclerotic renal artery stenosis will be tested in this study. The intervention group will be treated with paclitaxel eluting balloon. The control group will be treated with plain old balloon(POB). The primary endpoint is efficacy of blood pressure control.

DETAILED DESCRIPTION:
Renal artery stenosis is common cause for hypertension in young people. It could be treated with open surgery or endovascular intervention. Open surgery has relatively high complication rate. Endovascular intervention is micro-invasive but with high restenosis rate. Drug eluting balloon(DEB) has been demonstrated to be effective for preventing restenosis in peripheral arteries. This study aims to test the efficacy of drug eluting balloon for non-atherosclerotic renal artery stenosis. The intervention group will be treated with paclitaxel eluting balloon. The control group will be treated with plain old balloon. The primary endpoint is efficacy of blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18y and 45y.
2. with ≥ 60% stenosis in at least one renal artery.
3. with hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg).
4. patients with no severe renal insufficiency (eGFR>30 ml/min, length of the kidney ≥ 7cm).
5. Good compliance.
6. with informed consent.

Exclusion Criteria:

1. With apparent atherosclerotic risk factors.
2. With renal intervention or surgery history.
3. With congenital anatomical anomaly.
4. With severe renal insufficiency (length of the target kidney < 7cm, total eGFR<30ml/min, divided eGFR of the target kidney<8 ml/min)
5. With contraindication for antiplatelet therapy.
6. With severe cardiopulmonary insufficiency.
7. Allergic to contrast medium
8. Being pregnant or preparing for pregnancy
9. With active cancer.
10. Life expectancy < 12 month
11. Without informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate(cure or improvement of hypertension) | 9 months
  Cure: diastolic blood pressure <90 mm Hg and systolic blood pressure <140 mm Hg off antihypertensive medications. Improvement: diastolic blood pressure <90 mm Hg and/or systolic blood pressure <140 mm Hg on the same or reduced number of medications (or reduced number of defined daily doses as described by the World Health Organization ) or a reduction in diastolic blood pressure by at least 15 mm Hg on the same or reduced number of medications
Primary patency rate | 9 months
  uninterrupted patency with no procedures performed on or at the margins of the treated segment or bypass

SECONDARY OUTCOMES:
Technical success rate | immediately after intervention
  No residual stenosis more than 50%
complication rate | within 30 days post-intervention
  All complications occurring within 30 days or during the same hospitalization as the revascularization procedure
Bail-out stenting rate | during the procedure
  Stent implanted after angioplasty for residual stenosis of dissection
Clinical benefit rate | 1, 3,6,12 months
primary patency rate | 6,12 months
Renal function | 6,9,12 months
  eGFR (ml/min)
Renal function | 6,9,12 months
  serum Cr
secondary patency rate | 9, 12 months
  any procedure that restores patency after occlusion
Target lesion revascularization | 9,12 months
  either repeat percutaneous or surgical revascularization for a lesion anywhere within the angioplasty region or the 5-mm borders proximal or distal to angioplasty region

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Zheng, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No